CLINICAL TRIAL: NCT03439982
Title: A Prospective Single Center Open Label Trial of RBX2660 (Microbiota Suspension) in the Management of Hepatic Encephalopathy
Brief Title: Fecal Transplant for Hepatic Encephalopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Rebiotix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00060782
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2021-07

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic encephalopathy, fecal microbiota transplant
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT (Experimental): Open label FMT administered at week 0 by colonoscopy and weeks 1-4 by enema
  Interventions: Biological: FMT

INTERVENTIONS:
Biological: FMT — FMT processed from routinely screened donors

SUMMARY:
The purpose of the study is to determine if fecal microbiota transplant (FMT) can reverse hepatic encephalopathy (HE) in cirrhotic patients who continue to have breakthrough episodes of HE despite maintenance therapy with lactulose and/or rifaximin or metronidazole.

DETAILED DESCRIPTION:
Subjects receive FMT from a single donor by colonoscopy at week 0 and by enema at weeks 1-4. HE is measured by Inhibitory Control Test (ICT) and Stroop test as well as fasting serum ammonia levels.

ELIGIBILITY:
Inclusion Criteria:

* Adult cirrhotic patients of various etiology on lactulose and/pr rifaximin or metronidazole for minimum 4 weeks as secondary prophylaxis
* Abnormal ICT (>5 lures) or abnormal Stroop test (>200 seconds)
* Baseline Conn score 0 or 1
* Infectious etiology of HE has been ruled out

Exclusion Criteria:

* those with tense ascites
* those who do not provide assent
* life expectancy <3 months
* TIPS within the past 3 months
* neurologic disease such as dementia, Parkinson's, structural brain lesions
* pregnancy
* intestinal obstruction
* alcoholic hepatitis
* active alcohol or substance abuse
* those without stable social support
* concurrent infection such as spontaneous bacterial peritonitis, pneumonia or urinary tract infection
* creatinine clearance less that 50% compared to baseline
* hospital admission for HE within one month of enrollment
* active hepatocellular carcinoma
* active GI bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Portion of participants with normalization of ICT or Stroop Test during the study | 8 weeks

SECONDARY OUTCOMES:
Proportion of patients with normalization ICT or Stroop test scores at 1 week, 2 weeks, 4 weeks and 8 | 8 weeks
Changes in serum ammonia level pre and post FMT | 8 weeks
Changes in Quality of Life measured by Chronic Liver Disease Questionnaire (CDLQ) pre and post FMT | 8 weeks
  29 Questions Total- each question is on a seven point scales, ranging from the worst (1) to the best (7) possible function
Change in Intestinal Microbiota pre-and post FMT | 8 weeks
Serious Adverse Events | 8 weeks
  i) All serious adverse events up to and including week 8. A serious adverse event is any event which results in any of the following: i) Death ii) Colonic perforation iii) Proven infections as defined by the presence of i) spontaneous bacteremia: positive blood cultures in the absence of any other potential source of infection; ii) spontaneous bacterial peritonitis: ascetic fluid PMN equal to or greater than 250/mm3; iii) UTI: urinary leukocyte count greater than 15 cells per HPF and positive urine culture; vi) other infections identified by clinical, radiologic and bacteriologic results.
  iv) Possible infections as defined by i) fever (temp > 37.80 C), ii) leukocytosis (>15,000 mm3) or increased immature neutrophils in blood (>500 mm3), negative cultures and no other signs of infection.
Change in stool Bile Acids Composition pre and post FMT | 8 Weeks
Changes in stool short chain free fatty acids pre and post FMT | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — Associate Professor
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pun CK, Huang HC, Chang CC, Hsu SJ, Huang YH, Hou MC, Lee FY. Hepatic encephalopathy: From novel pathogenesis mechanism to emerging treatments. J Chin Med Assoc. 2024 Mar 1;87(3):245-251. doi: 10.1097/JCMA.0000000000001041. Epub 2023 Dec 18. PMID 38109364